CLINICAL TRIAL: NCT02472340
Title: Assessment and Reproducibility of Mitochondrial Function and Mitophagy Measurements in Human Muscle Tissue of Active and Pre Frail Elderly Males
Brief Title: Mitophagy and Autophagy in Elderly Subjects
Status: Completed | Type: Observational
Sponsor: Amazentis SA (Industry)
Collaborators: Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: CHDR1510; 15.01.AMZ (Other: Amazentis)
Record Dates: First submitted 2015-06-09; First posted 2015-06-15 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-03

CONDITIONS: Aging; Frailty; Mitophagy
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Muscle, Peripheral blood mononuclear cells (PBMC)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sedentary, Pre-frail: 10 sedentary, pre-frail elderly, >61 year of age
  Interventions: Procedure: Muscle Biopsy
- Active, Healthy: 10 Active, healthy elderly, >61 years of age
  Interventions: Procedure: Muscle Biopsy

INTERVENTIONS:
Procedure: Muscle Biopsy — Muscle Biopsy

SUMMARY:
In recent years, evidence has shown that mitochondrial dysfunction plays an important role in the development of age-related muscle decline that may lead to frailty.

During aging, there is a progressive reduction in the cell's capacity to eliminate its dysfunctional elements by autophagy, as evidenced by the accumulation of oxidative damage and mutations in mitochondria and by the decrease in autophagic flux. In fact, it has been demonstrated that dysfunctional mitochondria can be specifically targeted for elimination by autophagy, a process that has been termed mitophagy.

A major challenge in the clinic today is in the lack of validated tools, including biomarkers, to assess the decline in mitochondrial health associated with an impairment in muscle function. In the present study, the investigators will employ a battery of established and exploratory tests (clinical, physiological and molecular) to assess in vivo mitochondrial function and more specifically, the levels of mitophagy and autophagy, in the muscle of healthy and pre-frail elderly.

It is anticipated that the results of this study will facilitate the rapid translation of interventions targeting mitophagy and autophagy for the improvement of muscle function.

ELIGIBILITY:
Inclusion Criteria:

* for Active, Healthy subjects:

  1. >61 years of age, inclusive.
  2. Healthy male subjects. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, haematology, blood chemistry, and urinalysis.
  3. Body mass index (BMI) between 15 and 32 kg/m2, inclusive.
  4. Able to participate and willing to give written informed consent and to comply with the study restrictions.
  5. Category 2 or 3 as assessed by the International Physical Activity Questionnaires (IPAQ). Activity level is ≥ 600 MET (metabolic equivalent unit) - minutes per week.
  6. Normal physical performance: normal gait speed, i.e. a walking ≥ 0.8 m/s in the 4-m walking test.
  7. Normal muscle mass: normal skeletal muscle mass index (SMI), measured by Bioimpedance analysis (BIA, ≥ 10.75 kg/m2).
  8. Normal muscle strength: handgrip strength (measured with the Jamar dynamometer) of ≥ 30 kg.

for Sedentary, Pre-frail subjects:

1. Sedentary, pre-frail males. Pre-frailty is defined as fulfilling to at least two out of the following three criteria: low physical performance (low gait speed, i.e. a walking speed below 0.8 m/s in the 4-m walking test), low muscle mass (a low skeletal muscle mass index (SMI), measured by Bioimpedance analysis (BIA, < 10.75 kg/m2)) and/or low muscle strength: handgrip strength (measured with the Jamar dynamometer) of < 30 kg. Sedentary behaviour is defined as having an activity category of 1 as assessed by the International Physical Activity Questionnaires (IPAQ) (Activity level is ≥ 600 MET (metabolic equivalent unit) - minutes per week).
2. Body mass index (BMI) between 15 and 32 kg/m2, inclusive.
3. Able to participate and willing to give written informed consent and to comply with the study restrictions.
4. >61 years of age, inclusive.

Exclusion Criteria:

* for Active, Healthy subjects:

  1. Presence of any contraindication to have MRI scans performed (e.g. pacemaker, intracranial clips etc.).
  2. Having diabetes mellitus or lower extremity peripheral vascular disease, as these conditions may interfere with interpretation of the dynamic 31P-MRS and NIRS of the lower extremity.
  3. Participation in a clinical trial within 90 days of screening or more than 4 times in the previous year.
  4. A history (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol).
  5. Smoking within 3 months prior to screening and inability to refrain from smoking during the course of the study (from screening to End-of-Study [EOS]).
  6. A history or presence of allergy to 5-aminolevulinic acid or porphyrins.
  7. A history or presence of allergy to lidocaine.
  8. Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening.
  9. Loss or donation of blood over 500 mL within three months (males) or four months (females) prior to screening.
  10. Unwillingness or inability to refrain from consuming alcohol within 48 hours before each visit until the end of that visit.
  11. Unwillingness or inability to refrain from consuming 8 or more units of xanthine containing beverages and foods per day during the entire study.
  12. Unwillingness or inability to refrain from consuming the following supplements: L-carnitine, creatine, Q10, vitamin A, niacin, folic acid, vitamin C, vitamin E and probiotic- foods and supplements at least two weeks before study enrolment.
  13. Unwillingness or inability to have a muscle biopsy performed.

For Sedentary, Pre-frail subjects

1. Presence of any contraindication to have MRI scans performed (e.g. pacemaker, intracranial clips etc.).
2. Having diabetes mellitus or lower extremity peripheral vascular disease, as these conditions may interfere with interpretation of the dynamic 31P-MRS and NIRS of the lower extremity.
3. Participation in a clinical trial within 90 days of screening or more than 4 times in the previous year.
4. A history (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol).
5. Smoking within 3 months prior to screening and inability to refrain from smoking during the course of the study (from screening to EOS).
6. A history or presence of allergy to 5-aminolevulinic acid or porphyrins.
7. A history or presence of allergy to lidocaine.
8. Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening.
9. Loss or donation of blood over 500 mL within three months (males) or four months (females) prior to screening.
10. Unwillingness or inability to refrain from consuming alcohol within 48 hours before each visit until the end of that visit.
11. Unwillingness or inability to refrain from consuming 8 or more units of xanthine containing beverages and foods per day during the entire study.
12. Unwillingness or inability to refrain from consuming the following supplements: L-carnitine, creatine, Q10, vitamin A, niacin, folic acid, vitamin C, vitamin E and probiotic- foods and supplements at least two weeks before study enrolment.
13. Unwillingness or inability to have a muscle biopsy performed.
14. Underlying chronic disease, which, in the opinion of the investigator would interfere with study participation or the validity of the measurements.
15. Unintentional weight loss ≤5% of usual body weight during the last 6 months.
16. Anorexia or anorexia-related symptoms

Ages: 61 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 10 active, healthy elderly, >61 years of age
  * 10 sedentary, pre-frail elderly, >61 years of age
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Gene and protein expression for autophagy and mitophagy biomarkers in muscle tissue | 9 months

SECONDARY OUTCOMES:
PCr recovery time (in seconds) measured by 31P-MRS (31-Phosphorus Magnetic Resonance Spectroscopy). | 9 months
mVO2 (in ml/min/100 ml) in muscle measured by NIRS (Near-infrared Spectroscopy) | 9 months
MitoPO2 (in mmHg) in the skin measured by PpIX-TSLT (Protoporphyrin IX - Triplet State Lifetime Technique). | 9 months
Hand grip strength (in kg) measured by the Jamar dynamometer. | 9 months
Peak muscle force of quadriceps measured by handheld dynamometry | 9 months
Postural stability (in mm sway) measured by body sway | 9 months
Level of activity, using the Vital Connect HealthPatch accelerometer | 9 months
Short physical performance battery (SPPB) test. | 9 months

OTHER OUTCOMES:
Ratio of mtDNA to nuDNA in muscle | 9 months
Gene and protein expression for mitophagy and autophagy in PBMC's | 9 months
Skeletal muscle subtype via histology | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Geert Jan Groeneveld, MD, PhD, Principal Investigator — CHDR; Anurag Singh, MD, PhD, Study Director — Amazentis SA
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands